CLINICAL TRIAL: NCT00820859
Title: Treatment of Agitation in the Nursing Home
Brief Title: Treatment Routes for Exploring Agitation
Acronym: TREA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Jiska Cohen-Mansfield, Ph.D., Director, Research Institute on Aging
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IA0144; 5R01AG010172-11 (NIH)
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Dementia; Behavior Problems
Keywords: Cognition disorder; nursing home residents; agitation; behavior disorder
MeSH Terms: conditions — Dementia; Mental Disorders; Cognition Disorders; Psychomotor Agitation | interventions — Trehalase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: TREA (Treatment Routes for Exploring Agitation)
- 2 (Active Comparator)
  Interventions: Behavioral: Placebo Control Group

INTERVENTIONS:
Behavioral: TREA (Treatment Routes for Exploring Agitation) — Individualized non-pharmacological treatment plan for agitation
  Arms: 1
Behavioral: Placebo Control Group — A presentation on the treatment of behavior problems in dementia given to the staff caregivers of the comparison group
  Arms: 2

SUMMARY:
The purpose of this study is to examine the efficacy of non-pharmacological ways to treat agitated behaviors in nursing home residents with dementia. The hypothesis is that non-pharmacological interventions will be more effective than placebo in decreasing such behaviors.

DETAILED DESCRIPTION:
Clinicians often refer to elderly persons under their care as "agitated." However, agitation is not a diagnosis, but rather, a descriptive term pertaining to a group of behavioral signs and symptoms, defined as socially inappropriate verbal, vocal, or motor (physical) activity that is not judged by an outside observer to result directly from the needs or confusion of the agitated individual. While the literature reports positive effects of non-pharmacological interventions, most studies tend to be based on small samples and do not yield statistically significant results. This study examines the impact of non-pharmacologic interventions tailored through an algorithm labeled TREA (Treatment Routes for Exploring Agitation) using a large, well-controlled, systematic research design.

TREA is an objective, systematic method for developing individualized non-pharmacological treatment plans based on an analysis of the agitated person's unmet needs, past and current preferences, past role-identity, cognitive, mobility, and sensory abilities/limitations, and possible causes for particular agitated behaviors. The methodology calls for ascertaining the type of agitated behavior and the most likely etiology, and then matching the intervention to the etiology and to the participant's characteristics.

The protocol involves the following steps:

* Baseline assessment - using standardized assessments (e.g., MMSE, ABMI, CMAI, Self-identity in dementia), collecting background demographic and medical information as well as systematic observations of the agitated resident
* Intervention exploration - after analyzing potential unmet needs as well as preferences, abilities and identities of each participant, investigators develop a list of potentially successful interventions, examining the effectiveness of a wide range of interventions, from family videos to manipulatives (e.g., puzzles, a tool kit)
* Intervention (treatment) phase - Interventions are systematically provided during the hours of highest agitation (determined at baseline) and observations are conducted at the same time. The treatment phase lasts for 10 days. The placebo control group includes a presentation to staff members as to how to intervene with behavior problems and similar observations of residents.
* Follow-up phase includes repeated assessments without interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Diagnosis of dementia derived from the resident's medical chart at the facility or from an attending physician, as based on DSM-IV criteria and the Report of the NINCDS-ADRDA
* Resident of the facility for at least three weeks so that nursing staff members know the resident well enough to accurately assess him or her
* Identified by nursing staff to exhibit either verbal agitation or physical non-aggressive agitation at least several times a day

Exclusion Criteria:

* Lifelong diagnosis of schizophrenia
* Bipolar disorder diagnosed prior to onset of dementia
* Diagnosis of premorbid mental retardation
* Judged by direct-care nursing staff to have a life expectancy of less than 3 months
* Expected to leave the nursing home (either to enter the hospital or to go home) within the next 4 months
* Agitation manifested less than 6 times a day

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Agitation Behavior Mapping Instrument (ABMI) | 10 days of intervention vs. 10 days of baseline

SECONDARY OUTCOMES:
affect/mood measured by Lawton's behavior stream assessment | 10 days of intervention vs. 10 days of baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jiska Cohen-Mansfield, PhD, Principal Investigator — Research Institute on Aging
Locations (1):
- Research Institute on Aging, Rockville, Maryland, United States

REFERENCES:
- [Background] Cohen-Mansfield J. Agitated behavior in persons with dementia: the relationship between type of behavior, its frequency, and its disruptiveness. J Psychiatr Res. 2008 Nov;43(1):64-9. doi: 10.1016/j.jpsychires.2008.02.003. Epub 2008 Apr 3. PMID 18394647
- [Background] Cohen-Mansfield J, Libin A, Marx MS. Nonpharmacological treatment of agitation: a controlled trial of systematic individualized intervention. J Gerontol A Biol Sci Med Sci. 2007 Aug;62(8):908-16. doi: 10.1093/gerona/62.8.908. PMID 17702884
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Derived] Cohen-Mansfield J, Thein K, Marx MS, Dakheel-Ali M, Freedman L. Efficacy of nonpharmacologic interventions for agitation in advanced dementia: a randomized, placebo-controlled trial. J Clin Psychiatry. 2012 Sep;73(9):1255-61. doi: 10.4088/JCP.12m07918. PMID 23059151
- See also: Research Institute on Aging — http://www.researchinstituteonaging.org/